CLINICAL TRIAL: NCT04125381
Title: Chronic Exposure to Arsenic and Risk of Lung Cancer Among Residents in the Province of Viterbo, Central Italy.
Brief Title: Arsenic Exposure and Lung Cancer Incidence
Status: Completed | Type: Observational
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Leonardo Palombi, Leonardo Palombi, Full Professor of Hygiene and Preventive Medicine, University of Rome Tor Vergata
Other Study IDs: ArsenicVT2019
Record Dates: First submitted 2019-10-11; First posted 2019-10-14 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Incident Cases of Lung Cancer (Code ICD-O C340-C349)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed to high Arsenic concentration: All the inhabitants, residing in one of the municipalities of Viterbo Province with high Arsenic concentration in drinking water, were enrolled
  Interventions: Other: Exposure to Arsenic by drinking water
- Exposed to low Arsenic concentration: All the inhabitants, residing in one of the municipalities of Viterbo Province with low Arsenic concentration in drinking water, were enrolled
  Interventions: Other: Exposure to Arsenic by drinking water

INTERVENTIONS:
Other: Exposure to Arsenic by drinking water — People residing in municipalities with Arsenic drinking water concentrations over legal threshold (10 µg/L), were considered as exposed.

SUMMARY:
Aim of the study was to assess any associations between chronic exposure by drinking water to Arsenic and onset of lung cancer, using a retrospective cohort study design.

Incident cases of lung cancer from 1st January 2006 to 31st December 2012, recorded by Viterbo Cancer Registry, occurring during the period, were considered as primary outcome. People residing in municipalities with Arsenic drinking water concentrations over legal threshold (10 µg/L) were considered as exposed.

DETAILED DESCRIPTION:
Arsenic and its compounds were classified as human carcinogens by IARC, because of their role in the onset and the progression of several neoplasms: liver, lung, bladder, prostate and skin cancer. If many studies shed to light on the existence of a strong association between As and cancer at chronic exposure to high metalloid concentrations (>150 µg/L), much remains to be clarified on the effects of low-moderate exposure, such as those occurring in Italy. The aim of this retrospective cohort study is to focus on the role of Arsenic in the pathogenesis of lung cancer, as one of the most impacting neoplasms in terms of incidence and prevalence (40.000 new diagnoses in Italy in 2017), in Viterbo Province, central Italy.

Because of its high toxicity and its ubiquitous distribution, that earned the metalloid the first in the Priority list by ATSDR, thus being a main issue in Public Health.

Materials and Methods From 1st January 2006 to 31st December 2012 all the inhabitants, residing in one of the 60 municipalities of Viterbo Province (around 320,279 people) were enrolled. Incident cases of lung cancer, recorded by Viterbo Cancer Registry, occurring during the period, were considered as primary outcome. People residing in municipalities with Arsenic drinking water concentrations over legal threshold (10 µg/L), as provided by Arpa Lazio, were considered as exposed.

Risk difference in developing lung cancer among exposed and not exposed was estimated by Relative Risk (RR) and Attributable Risk (AR).

ELIGIBILITY:
Inclusion Criteria:

From 1st January 2006 to 31st December 2012 all the inhabitants, residing in one of the 60 municipalities of Viterbo Province were enrolled.

Exclusion Criteria:

No exclusion criteria were applied

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All the residents of the Viterbo Province, Central Italy
Sampling Method: Non-Probability Sample
Enrollment: 314000 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-03-18 (Actual)

PRIMARY OUTCOMES:
Incident cases of lung cancer | 2006-2012
  Incident cases of lung cancer (code ICDO C340-C349), recorded by Viterbo Cancer Registry

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Palombi, MD, Principal Investigator — University Rome Tor Vergata, Roma (Italy)
Locations (1):
- Cancer Registry Viterbo Province, Viterbo, Italy

IPD SHARING:
Plan to Share IPD: Undecided